CLINICAL TRIAL: NCT02678741
Title: Multi-center Phase I/IIa Trial of an Autologous Tumor Lysate (TL) + Yeast Cell Wall Particles (YCWP) + Dendritic Cells (DC) Vaccine in Addition to Standard of Care Checkpoint Inhibitor of Choice in Metastatic Melanoma Patients With Measurable Disease.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Elios Therapeutics, LLC (Industry)
Collaborators: LumaBridge (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20152397
Record Dates: First submitted 2016-02-04; First posted 2016-02-10 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No clinical response (Active Comparator): No clinical response (PD de novo) after a minimum of 3 months on CPI monotherapy
  Interventions: Drug: TLPLDC Vaccine
- Develop PD (Active Comparator): Develop PD after initial clinical response to CPI monotherapy
  Interventions: Drug: TLPLDC Vaccine
- Stable Disease (Active Comparator): Stable disease for at least 6 months on CPI monotherapy
  Interventions: Drug: TLPLDC Vaccine

INTERVENTIONS:
Drug: TLPLDC Vaccine — Tumor Lysate, Particle Loaded, Dendritic Cell Vaccine

SUMMARY:
Assess the safety and tumor response of utilizing an autologous tumor lysate, particle-loaded, dendritic cell (TLPLDC) vaccine given in combination with standard of care (SoC) checkpoint inhibitors (CPI) in patients with stage IV melanoma with measurable disease.

DETAILED DESCRIPTION:
Metastatic melanoma patients eligible for (or currently on) CPI therapy per SoC will be identified and screened for inclusion/exclusion criteria. Eligible patients will be counseled and consented for tissue procurement. They will undergo excisional or core needle biopsy as clinically indicated and this tissue will be shipped in liquid nitrogen shippers through FedEx to our central facility in Greenville, SC.The tumor will be stored frozen until vaccine preparation. Vaccine development requires 48 hours for preparation. Upon verification that adequate tissue was obtained, these patients will then be counseled and consented for participation in the trial.

The patients who qualify for participation in this trial will continue their treatment of CPI. Once consented, patients will receive a single injection of Neupogen (G-CSF) 300 μg SQ 24-48 hrs prior to having 70 mL of blood collected and sent to our central facility for DC isolation and preparation. Those who cannot tolerate Neupogen or refuse it will have 120 mL of blood drawn and sent. Additional blood may be drawn if additional vaccine doses need to be made or re-made for any reason. Vaccines will be prepared by producing TL through freeze/thaw cycling and then loaded into pre-prepared YCWP. The TL-loaded YCWP will be introduced to the DC for phagocytosis thus creating the TLPLDC vaccine, which will be frozen in single dose vials. Each vial will contain 1 x 106 TLPLDC and will be labeled with the patient's unique study number.

The frozen autologous TLPLDC will be sent back to the site with a total of 6 single dose vials after the vaccine has completed QA/QC testing and lot-release (usually 3 weeks). The primary vaccination series will include monthly inoculations at 0, 1, 2, 3 months followed by boosters at 6 and 9 months in the same lymph node draining area (preferably the anterior thigh). Once received, the first inoculation should occur within 4 weeks.

Safety data will be collected on local and systemic toxicities and graded and reported per the Common Terminology Criteria for Adverse Events (CTCAE) v4.03.

Patients will follow-up at their respective sites for evaluation of metastatic disease per SoC. They will under imaging, CT/PET-CT, to meet Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 and iRECIST to monitor disease.

Blood (50 mL) will be collected from all patients prior to each inoculation and at 12 months from enrollment for a total of 7 time points or a total of 350 mL of blood over 1 year. The collected blood will be sent to our central facility for immunologic testing of T-cell responses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Appendix A)
* Metastatic melanoma eligible for {or currently on} standard of care CPI therapy (treating physician's choice) with measurable disease.
* Approximately 1 cm3 preferred but 1 mg minimum of accessible and dispensable tumor (minimum of 3 passes with a core needle)
* Able to tolerate CPI treatment regimen {if already started}
* Adequate organ function as determined by the following laboratory values:
* ANC ≥ 1,000/μL
* Platelets ≥ 75,000/μL
* Hgb ≥ 9 g/dL
* Creatinine ≤ 1.5 x upper limit of normal (ULN) or Creatinine clearance ≥ 50% of lower limit of normal (LLN)
* Total bilirubin ≤ 1.5 ULN
* ALT and AST ≤ 1.5 ULN
* For women of child-bearing potential, agreement to use adequate birth control (abstinence, hysterectomy, bilateral oophorectomy, bilateral tubal ligation, oral contraception, IUD, or use of condoms or diaphragms)

Exclusion Criteria:

* Inability to tolerate CPI therapy {if already started}
* Rapidly progressing multi-focal metastatic melanoma
* Insufficient tumor available to produce vaccine
* ECOG >2 performance status (Appendix A)
* Immune deficiency disease or known history of HIV, HBV, HCV
* Receiving immunosuppressive therapy including chronic steroids (except physiologic maintenance doses), methotrexate, or other known immunosuppressive agents
* Pregnancy (assessed by urine HCG)
* Breast feeding
* Active pulmonary disease requiring medication to include multiple inhalers (>2 inhalers and one containing steroids)
* Involved in other experimental protocols (except with permission of the other study PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02; Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Peoples, MD, Study Director — LumaBridge
Locations (7):
- United States (7):
  - University of Alabama Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - John Wayne Cancer Institute/Providence Saint John's Health Center, Santa Monica, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Northside Hospital, Atlanta, Georgia
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Providence Regional Medical Center, Everett, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrollees evaluated across all arms.
Groups:
- Treatment Group: TLPLDC Vaccine: Tumor Lysate, Particle Loaded, Dendritic Cell Vaccine
Period: Overall Study
Arm/Group | Treatment Group
Started | 26
No Clinical Response | 3
Stable Disease | 2
Progressive Disease | 10
Completed | 6
Not Completed | 20
Not completed — Death | 4
Not completed — Withdrawal by Subject | 1
Not completed — ineligible | 3
Not completed — Not RECIST Measurable | 2
Not completed — Lack of Efficacy | 10

BASELINE CHARACTERISTICS:
Groups:
- Treatment: TLPLDC Vaccine: Tumor Lysate, Particle Loaded, Dendritic Cell Vaccine
Arm/Group | Treatment
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Graded Standard Systemic Toxicities (Using CTCAE Graded Toxicity Scale) by Patient
Description: Safety of adding the TLPLDC vaccine to SoC CPI monotherapy
Time Frame: 12 months (1 year)
Population: The safety evaluation of TLPLDC was the primary endpoint of this phase 1 trial. There were 26 patients enrolled, and 16 received at least one dose of vaccine. The population used for the safety analysis included these 16 patients. Toxicity was graded per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
  A total of 60 inoculations of TLPLDC were given to 16 patients, with the median of 3.5 inoculations.
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 16
participants | 12

2. Primary Outcome: Graded Standard Systemic Toxicities (Using CTCAE Graded Toxicity Scale) by Number of AEs
Description: Safety of adding the TLPLDC vaccine to SoC CPI monotherapy
Time Frame: 12 months (1 year)
Measure: Number; unit: events
Arm/Group | Treatment
Number analyzed (Participants) | 16
events
  AEs related to TLPLDC | 12
  Total AEs | 79
  Serious AEs or Deaths | 0

3. Secondary Outcome: Tumor Response to Treatment Using Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: RECIST criteria is used for assessing tumor response in the addition of TLPLDC vaccine. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 12 months (1 year)
Population: Of 26 patients enrolled, 16 received at least one inoculation with the TLPLDC vaccine; The 16 patients who received at least one inoculation were included in the efficacy analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 16
Participants
  No Clinical Response | 2
  Progressive Disease | 10
  Stable Disease | 2
  Not RECIST evaluable | 2

ADVERSE EVENTS:
Time Frame: Safety data was collected on local and systemic toxicities, graded and reported per the NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.03 (Appendix C) (7). Patients followed up at their respective sites for evaluation of metastatic disease per NCCN guidelines (2)]. Patients underwent imaging to monitor disease approximately every 3 months for 1 year.
Description: Imaging was done with the same modality that was used for baseline measurements, to meet RECIST criteria (5) Time to the best overall response was determined from the date of first inoculation until the first day that the tumor meets RECIST criteria for a particular tumor response
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 4/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 12/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=16)
Syncope (Cardiac disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1)
Injection site rxn (Skin and subcutaneous tissue disorders) | 1 (1)
skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT02678741/Prot_SAP_000.pdf